CLINICAL TRIAL: NCT06126354
Title: Role of Hyperinsulinemia in NAFLD: Dexamethasone-Pancreatic Clamp Pilot & Feasibility Study
Brief Title: Dexamethasone/Pancreatic Clamp P&F
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigators' scientific priorities shifted.
Sponsor: Columbia University (Other)
Collaborators: Albert Einstein College of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAU7680; 3P30DK063608 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Insulin Resistance; Prediabetic State; Non-Alcoholic Fatty Liver Disease; Overweight and Obesity
Keywords: Insulin resistance; Hyperinsulinemia; Diabetes; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Non-alcoholic Fatty Liver Disease; Overweight; Obesity; Hyperinsulinism; Diabetes Mellitus | interventions — Insulin; Octreotide; Glucagon; Human Growth Hormone; Dexamethasone; Glucose; Saline Solution; Serum Albumin, Human

STUDY DESIGN:
Intervention Model Description: All participants will undergo (i.e., cross over between) both pancreatic clamp protocols (MH, RE) separated by 2-4 weeks. The order of the clamp protocols (i.e., MH > RE, RE > MH) will be randomized.
Who Masked: Participant
Masking Description: Participant will be blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance hyperinsulinemia (MH) protocol (Active Comparator): The basal insulin infusion rate (IIR) necessary to maintain participants' mean basal fasting plasma glucose (mbFPG) will be determined during the basal titration period. Then, during the intervention period, the IIR will remain at 100% of basal for the full duration (225 min). The IIR and resulting insulin levels are expected to be relatively high (cf. hyperinsulinemia) because of dexamethasone-induced insulin resistance.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Human Growth Hormone; Drug: Dexamethasone Oral; Other: [6,6-2H2] D-glucose; Drug: 20% D-glucose (aq); Dietary Supplement: BOOST Plus; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer; Other: Normal saline; Other: Human albumin
- Reduction toward euinsulinemia (RE) protocol (Experimental): The basal insulin infusion rate (IIR) necessary to maintain participants' mean basal fasting plasma glucose (mbFPG) will be determined during the basal titration period. Then, during the intervention period, the IIR will be reduced progressively, at 75-min intervals, to 90%, 75%, and 60% of basal IIR. Thus, the basal hyperinsulinemia expected due to underlying insulin resistance will be reduced toward euinsulinemia.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Human Growth Hormone; Drug: Dexamethasone Oral; Other: [6,6-2H2] D-glucose; Drug: 20% D-glucose (aq); Dietary Supplement: BOOST Plus; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer; Other: Normal saline; Other: Human albumin

INTERVENTIONS:
Drug: Insulin human — Insulin infusion rate (IIR) will be determined empirically first to maintain mean basal fasting plasma glucose, and then either maintained at the basal rate (MH protocol) or be reduced stepwise toward euinsulinemia (RE protocol).
  Other Names: Novolin-R; Humulin-R
Drug: Octreotide Acetate — Octreotide will be infused at 30 ng/kg/min to suppress endogenous insulin, glucagon, and growth hormone secretion. Co-administered with glucagon and rhGH.
  Other Names: Octreotide Acetate IV
Drug: Glucagon — Glucagon will be replaced at a constant rate of up to 0.65 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and rhGH.
  Other Names: Glucagon IV
Drug: Human Growth Hormone — Recombinant human growth hormone (rhGH) will be replaced at a constant rate of up to 3 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and glucagon.
  Other Names: Omnitrope
Drug: Dexamethasone Oral — Synthetic pure glucocorticoid used to induce temporary insulin resistance, administered orally as seven 1-mg doses over 72 hours.
  Other Names: Dexamethasone
Other: [6,6-2H2] D-glucose — Stable isotope tracer administered to calculate glucose kinetics during pancreatic clamp.
  (Non-investigational)
  Other Names: D2-glucose, D2G
Drug: 20% D-glucose (aq) — 20% D-glucose (aq) (D20W) will be administered to counteract hypoglycemia or strongly downward blood glucose trends, as needed.
  (Non-investigational)
  Other Names: D20W
Dietary Supplement: BOOST Plus — Nutritional supplement will be administered to provide three standardized "mixed meals" on the day before the pancreatic clamp.
  (Non-investigational)
Device: Harvard Apparatus PHD ULTRA CP syringe pump — Device: Harvard Apparatus PHD ULTRA CP syringe pump Syringe pump used for highly precise administration of insulin, octreotide/glucagon/rhGH, and D20W (as needed) even at low infusion rates.
  (Non-investigational)
Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer — Glucose oxidase analyzer used to detect plasma glucose levels at the point of care. YSI have been the gold standard in clamp studies for many years. Two machines will run in parallel to ensure accuracy of results.
  (Non-investigational)
Other: Normal saline — Normal saline (0.9% NaCl, aq), variable rate (as needed)
  Other Names: NaCl IV
Other: Human albumin — Human albumin (5%, aq), 0.4 g per 100 mL of infusion (0.4% (w/v) in insulin and OCT/GCG/GH bags)
  Other Names: Human albumin IV

SUMMARY:
This is a single-center, prospective, randomized, controlled (crossover) clinical study designed to investigate the specific dose-response impact of insulin infusion rate (IIR) on blood glucose levels during a pancreatic clamp study in the setting of dexamethasone-induced insulin resistance. The investigators will recruit participants with a history of overweight/obesity but no history of prediabetes or diabetes. Participants will be rendered temporarily insulin resistant by taking seven doses of dexamethasone. They will then undergo two pancreatic clamp procedures in which individualized basal IIR are identified, followed in one by maintenance of basal IIR (maintenance hyperinsulinemia, MH) and in the other by a stepped decline in IIR (reduction toward euinsulinemia, RE). In both clamps the investigators will closely monitor plasma glucose and various metabolic parameters. The primary outcome will be the absolute and relative changes in steady-state plasma glucose levels at each stepped decline in IIR.

DETAILED DESCRIPTION:
Although high blood sugar and risk of heart disease are the most well-known health effects of type 2 diabetes (T2DM), nonalcoholic fatty liver disease (NAFLD), in which too much fat accumulates in the liver, has come to be recognized as another important complication. Unchecked, NAFLD can progress to severe liver inflammation, liver failure, and even liver cancer. The investigators suspect that high levels of the blood sugar-lowering hormone insulin leads to excessive fat production by the liver, and so lowering insulin levels might help to improve NAFLD. In order to answer this question, the investigators will temporarily render volunteers insulin resistant -- that is, simulating the risk of T2DM and NAFLD -- using seven doses of dexamethasone. They will then perform a "pancreatic clamp" - a procedure in which the body's production of insulin is temporarily shut off and then replaced at the same or lower levels. Again, the investigators expect that lowering insulin levels will lower fat production. Because this is a new research approach, the investigators first need to understand how lowering insulin levels affects blood sugar. Research participants in this pilot study will therefore undergo two pancreatic clamps, each following seven doses of dexamethasone, in random order: one roughly maintaining their own internal ("basal") insulin level and one in which the investigators lower that basal insulin level by 10%, 20%, and 40%. In each case, the investigators will observe the absolute and relative changes in blood sugar and the levels of certain fats as the investigators change the insulin level. Once the investigators have found a lower insulin level that they can safely maintain, the investigators will go on to study its effect on fat production in a later study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (using highly effective contraception if of childbearing potential) aged 18-65 years
2. Body mass index of 25.0-39.9 kg/m2
3. Able to understand written and spoken English and/or Spanish
4. Evidence of normal glucose metabolism (euglycemia), represented by not meeting the American Diabetes Association's definitions for prediabetes, impaired fasting glucose (IFG), or diabetes on screening labs. Thus, participants must meet both of the following conditions on screening labs:

   i. Prediabetes: Hemoglobin A1c < 5.7% ii. IFG: plasma glucose of < 100 mg/dL after 8-h fast
5. Normal fasting serum insulin (fasting insulin level < 12 μIU/mL) on screening labs
6. Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Unable to provide informed consent in English or Spanish
2. Concerns arising at screening visit (any of the following):

   i. Unwillingness to use only bedpan or urinal to void or to refrain from non-emergent mobile device use during the clamp ii. Unwillingness to fast (except water) for up to 24 hours iii. Documented weight loss of ≥ 5% of baseline within the previous 6 months iv. Abnormal blood pressure (including on treatment, if prescribed)
   * Systolic blood pressure < 90 mm Hg or > 160 mm Hg, and/or
   * Diastolic blood pressure < 60 mm Hg or > 100 mm Hg v. Abnormal resting heart rate: < 60 or ≥100 bpm
   * Sinus brady- or tachycardia that has been extensively worked up and considered benign by the recruit's personal physician may be permitted at the PI's discretion vi. Abnormal screening electrocardiogram (or if on file, performed within previous 90 d):
   * Non-sinus rhythm
   * Significant QTc prolongation (≥ 480 ms)
   * New or previously unknown ischaemic changes that persist on repeat EKG: ST elevations, T-wave inversions vii. Laboratory evidence of impaired glucose metabolism:
   * Hemoglobin A1c ≥ 5.7%, and/or
   * Fasting plasma glucose ≥ 100 mg/dL viii. Positive qualitative human chorionic gonadotropin, beta subunit (β-hCG) in women of childbearing potential ix. Positive urine drug screen, except for lawfully prescribed medications and/or marijuana x. Liver function abnormalities (either of the following)
   * Transaminases (AST or ALT) > 2.0 x the upper limit of normal
   * Total bilirubin > 1.25 x the upper limit of normal xi. Abnormal fasting lipids at screening (either of the following)
   * Triglycerides ≥ 400 mg/dL
   * LDL-cholesterol ≥ 190 mg/dL xii. Abnormal screening serum electrolytes (any of the following)
   * Abnormal sodium, potassium, chloride, or bicarbonate levels that are considered potentially significant according to the clinical judgment of the PI.
   * Creatinine equating to estimated glomerular filtration rate < 60 mL/min/1.73 m2 xiii. Abnormal complete blood count (CBC) (any of the following)
   * Hemoglobin < 10 g/dL or hematocrit < 30%
   * Platelet count < 100,000/μL
   * Exempt from CBC requirement if previously obtained value within 2 months of screening is available
3. Unwillingness to comply with masking and COVID-19 testing requirements per hospital policy
4. Reproductive concerns i. Women of childbearing potential not using highly effective contraception, defined as:

   * Surgical sterilization (e.g., bilateral tubal occlusion, bilateral oophorectomy and/or salpingectomy, hysterectomy)
   * Oral contraceptive pills taken daily, including during the study
   * Intrauterine device (levonorgestrel-eluting or copper) active at the time of study
   * Medroxyprogesterone acetate (Depo-Provera®) injection active at the time of study
   * Etonogestrel implants (e.g., Implanon®, etc.) active at the time of the study
   * Etonogestrel/ethinyl estradiol vaginal ring (e.g., NuvaRing®, etc.) active at the time of the study
   * Norelgestromin/ethinyl estradiol transdermal system (e.g., Ortho-Evra®) active at the time of the study ii. Women currently pregnant, measured by serum and/or urine β-hCG iii. Women currently breastfeeding
5. Concerns related to glucose metabolism i. Known, documented history of having met any of the American Diabetes Association's definitions of prediabetic state or of diabetes mellitus (i.e., overt diabetes):

   * Hemoglobin A1c ≥ 5.7%

     o Or rapid rise in documented HbA1c values causing clinical concern for evolving insulin deficiency
   * Plasma glucose ≥ 100 mg/dL after 8-h fast
   * Plasma glucose of ≥ 140 mg/dL at 2 h after ingestion of a 75-g glucose load
   * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state ii. History of gestational diabetes mellitus within the previous 5 years iii. Use of most antidiabetic medications within the 90 days prior to screening
   * Excluded: thiazolidinediones, sulfonylureas, meglitinides, dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, sodium-glucose cotransporter-2 (SGLT2) inhibitors, amylin mimetics, acarbose, insulin
   * Metformin used for weight control or polycystic ovarian syndrome is acceptable provided that recruits meet all of the inclusion criteria at screening iv. Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease) v. Fasting plasma glucose < 70 mg/dL at screening
6. Concerns related to lipid metabolism i. Known diagnoses of familial hypercholesterolemia, familial combined hyperlipidemia, or familial hyperchylomicronemia in the participant or a first-degree relative ii. Use of certain lipid-lowering drugs within 90 d prior to screening visit:

   * Statins or PCSK9 inhibitors for secondary prevention or treatment of familial hypercholesterolemia

     o Statins or PCSK9 inhibitors for primary prevention of ASCVD are acceptable
   * Fibrates (e.g., fenofibrate, clofibrate, gemfibrozil)
   * High-dose niacin (>100 mg daily)
7. Known, documented history, at the time of screening, of any of the following medical conditions:

   i. Pancreatic pathology, including but not limited to:
   * Pancreatic neoplasia
   * Chronic pancreatitis
   * Acute pancreatitis (or history of within the past 5 years)
   * Autoimmune pancreatitis
   * Surgical removal of any portion of the pancreas ii. Cardiovascular diseases (N.B. uncomplicated hypertension is not exclusionary)
   * Atherosclerotic cardiovascular disease
   * Stable or unstable angina
   * Myocardial infarction
   * Ischaemic or hemorrhagic stroke
   * Peripheral arterial disease (claudication)
   * Use of dual antiplatelet therapy (aspirin + P2Y12 inhibitor) Heart rhythm abnormalities
   * Congestive heart failure of any New York Heart Association class
   * Severe valvular heart disease (e.g., aortic stenosis)
   * Pulmonary hypertension iii. Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL/min/1.73 m2), of any cause iv. Advanced or severe liver disease, including but not limited to:
   * Advanced liver fibrosis, as determined by non-invasive testing
   * Cirrhosis of any etiology
   * Autoimmune hepatitis or other rheumatologic disorder affecting the liver
   * Biliopathy (e.g., progressive sclerosing cholangitis, primary biliary cholangitis)
   * Chronic liver infection (e.g., viral hepatitis, parasitic infestation)
   * Hepatocellular carcinoma
   * Infiltrative disorders (e.g., sarcoidosis, hemochromatosis, Wilson disease) v. Gallstone disease, including:
   * Biliary colic (active)
   * History of acute cholecystitis not treated with cholecystectomy
   * History of other gallstone complications (e.g., pancreatitis, cholangitis) vi.Chronic viral illness (N.B. diagnosis based only on medical history; we will not test for any of these viruses at any point in this study)
   * Hepatitis B virus (HBV), unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 90 d prior to screening
   * Hepatitis C virus (HCV) infection, unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 90 d prior to screening
   * Human immunodeficiency virus (HIV) infection vii. Malabsorptive conditions (active)
   * Active inflammatory bowel disease (quiescent and off medication is acceptable)
   * Celiac disease (in remission with gluten-free diet is acceptable)
   * Surgical removal of a significant length of intestine viii. Active seizure disorder (including controlled with antiepileptic drugs) ix. Psychiatric diseases causing functional impairment that:
   * Are or have been decompensated within 1 year of screening, and/or
   * Require use of anti-dopaminergic antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine), monoamine oxidase inhibitors, or lithium x. Other endocrinopathies:
   * Cushing syndrome (okay if considered in remission after treatment, provided that no exogenous corticosteroids or other ongoing treatment are required)
   * Adrenal insufficiency
   * Primary aldosteronism xi. Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation xii. Bleeding disorders, including due to anticoagulation, or significant anemia (see above) xiii. Dysautonomia, including post-vagotomy xiv. Active malignancy, or hormonally active benign neoplasm, except allowances for:
   * Non-melanoma skin cancer
   * Differentiated thyroid cancer (AJCC Stage I only)
8. Clinical concern for increased risk of volume overload, including due to medications and/or heart/liver/kidney problems, as listed above
9. Clinical concern for increased risk of hypokalemia, including low potassium on screening labs (i.e., below lower limit of normal)
10. Use of certain medications currently or within 30 d prior to screening:

    i. Prescribed medications used for any of the indications in the preceding list (§5.3.7) of excluded conditions, or their use within 90 d prior to screening, except allowances for:

    • Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above (e.g., antiepileptic drugs used for non-seizure indications, angiotensin converting enzyme inhibitor [ACEi]/angiotensin receptor blocker [ARB] used for uncomplicated hypertension rather than for congestive heart failure, etc.)

    o Note, as above, that antidiabetic drugs except metformin within 90 d of screening are excluded ii. Oral or parenteral corticosteroids for more than 3 days within the previous 30 days; topical and inhaled formulations are permitted iii. Fludrocortisone iv. Beta blockers or non-dihydropyridine calcium channel blockers (verapamil or diltiazem)
11. History of certain weight-loss (bariatric) surgery, including:

    i. Roux-en-Y gastric bypass ii. Biliopancreatic diversion iii. Restrictive procedures (lap band, sleeve gastrectomy) performed within the past 6 months
12. Clinical concern for alcohol overuse, including recent documented history during screening and/or participant report of regularly consuming more than 2 drinks per day for males or 1 drink per day for females.
13. Positive urine drug screen, with exceptions for:

    * Lawfully prescribed medications
    * Marijuana/tetrahydrocannabinol positivity, provided that the participant agrees not to use it during the same period that they will abstain from alcohol)
14. History of severe infection or ongoing febrile illness within 30 days of screening
15. Any other disease, condition, or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
16. Known allergy/hypersensitivity to any component of the medicinal product formulations, foods (including soy, dairy, peanuts, tree nuts, or egg), IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
17. Concurrent enrollment in another clinical study of any investigational drug therapy within 6 months prior to screening or within 5 half-lives of an investigational agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Absolute values of plasma glucose | Up to 425 minutes from the start of the procedure
  Goal is first to clamp insulin infusion rate to maintain mean basal fasting plasma glucose during the basal titration phase, and then during the intervention phase to observe the glucose levels that result from altering the basal IIR. Units: mg/dL
Relative change in plasma glucose | Up to 425 minutes from the start of the procedure
  Goal is first to clamp insulin infusion rate to maintain mean basal fasting plasma glucose during the basal titration phase, and then during the intervention phase to observe the impact of altering the basal IIR on glycemia. Units: fold difference and/or ∆mg/dL relative to previous time points
Absolute values of serum insulin | Up to 425 minutes from the start of the procedure
  Investigators will assess the insulin levels attained at the basal IIR, and at each stepwise reduction in IIR during the intervention phase. Units: micro-international units per milliliter (µIU/mL)
Relative change in serum insulin | Up to 425 minutes from the start of the procedure
  Investigators will compare the baseline insulin level to that attained at the basal IIR, as well as comparing to the change in insulin level that occurs with alterations in the IIR during the intervention phase. Units: fold difference and/or ∆ µIU/mL relative to previous time points
Absolute values of serum C-peptide | Up to 425 minutes from the start of the procedure
  Suppression of endogenous insulin by octreotide during pancreatic clamp is expected to result in a fall in C-peptide levels to near zero. Units: ng/mL
Relative change in serum C-peptide | Up to 425 minutes from the start of the procedure
  Suppression of endogenous insulin by octreotide during pancreatic clamp is expected to result in a fall in C-peptide levels to near zero. Units: fold difference and/or ∆ µIU/mL relative to previous time points

SECONDARY OUTCOMES:
Absolute values of serum or plasma triglyceride (TG) | Up to 425 minutes from the start of the procedure
  TG levels in serum reflect hepatic synthesis/storage and very low-density lipoprotein (VLDL) secretion. (units: mg/dL)
Relative change in absolute values of serum or plasma triglyceride (TG) | Up to 425 minutes from the start of the procedure
  TG levels in serum reflect hepatic synthesis/storage and VLDL secretion. (units: fold difference and/or ∆mg/dL relative to previous time points)
Absolute values of serum or plasma free fatty acid (FFA) | Up to 425 minutes from the start of the procedure
  FFA levels reflect adipose tissue lipolysis and its response to insulin and counterregulatory hormones. (units: mg/dL)
Relative change in serum or plasma free fatty acid (FFA) | Up to 425 minutes from the start of the procedure
  FFA levels reflect adipose tissue lipolysis and its response to insulin and counterregulatory hormones. (units: fold difference and/or ∆mg/dL relative to previous time points)
Absolute values of serum or plasma apolipoprotein B (ApoB) | Up to 425 minutes from the start of the procedure
  ApoB level is a surrogate for triglyceride-rich lipoproteins, especially hepatic VLDL. (units: mg/dL)
Relative change in serum or plasma apolipoprotein B (ApoB) | Up to 425 minutes from the start of the procedure
  ApoB level is a surrogate for triglyceride-rich lipoproteins, especially hepatic VLDL. (units: fold difference and/or ∆mg/dL relative to previous time points)
Plasma glucose kinetics: rate of appearance | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from [6,6-2H2] D-glucose (D2G) tracer enrichment by the Steele equations. (units: mg/kg/min)
Plasma glucose kinetics: rate of disappearance | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from D2G tracer enrichment by the Steele equations. (units: mg/kg/min)
Plasma glucose kinetics: endogenous glucose production | Measured every 5 minutes x 4 at the end of each steady-state IIR period, up to 425 minutes from the start of the procedure
  Calculated from D2G tracer enrichment by the Steele equations. (units: mg/kg/min)

OTHER OUTCOMES:
Absolute values of serum/plasma glucagon | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous glucagon replacement. (units: ng/L)
Relative change in serum or plasma glucagon | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous glucagon replacement. (units: fold difference and/or ∆ng/L relative to previous time points)
Absolute values of serum or plasma growth hormone | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous rhGH replacement. (units: ng/mL)
Relative change in serum or plasma growth hormone | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of exogenous rhGH replacement. (units: fold difference and/or ∆ng/mL relative to previous time points)
Serum cortisol level | Up to 425 minutes from the start of the procedure
  Assesses the adequacy of dexamethasone suppression of the hypothalamic-pituitary-adrenal axis. (units: μg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Blood samples will be banked in our Insulin Resistance Biobank and will be made available to other researchers for legitimate research purposes upon request. Associated data will be shared along with specimens in the smallest possible quantity and on a need-to-know basis. No Protected Health Information (PHI) will ever be disclosed to other researchers. All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of an Institutional Review Board-approved Material Transfer Agreement (MTA) and/or Data Use Agreement (DUA), as appropriate.
  IPD will be shared in a publicly accessible repository per NIH policy.
Supporting Information: Study Protocol
Time Frame: Indefinitely following study completion.
Access Criteria: All requests will be reviewed by the PI for scientific merit and samples/data will be transferred only upon completion of a MTA or DUA, as appropriate. No PHI will be disclosed or shared.